CLINICAL TRIAL: NCT00241527
Title: Efficacy of Esomeprazole 40 mg Once Daily Versus Placebo and Esomeprazole 20 mg Once Daily Versus Placebo in Treatment for Relief of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs Including COX-2 Selective NSAIDs
Brief Title: Esomeprazole for Relief of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9617C00003; SH-NEN-0003
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: NSAIDs; Upper GI Symptoms
MeSH Terms: interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
This study was a randomised, double-blind, parallel-group and placebo controlled study comparing the efficacy of esomeprazole 40 mg orally qd vs placebo and esomeprazole 20 mg orally qd vs placebo when given to patients on continuous use of NSAIDs, including COX-2 selective NSAIDs, for a treatment period of 4 weeks for relief of upper GI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* 18 years of age, or older.
* Capable of completing the diary card.
* Ability to complete the HRQL questionnaires.
* A clinical diagnosis of a chronic condition (e.g., osteoarthritis or rheumatoid arthritis) that requires continuous daily NSAID treatment for at least 7 months. Daily NSAID treatment is defined as taking the prescribed dose for at least 5 of 7 days in any given week and can include COX-2 selective NSAIDs, multiple NSAIDs, and high-dose aspirin (>325 mg/day).
* Daily NSAID treatment dose and type: (Must have been stable for at least 4 weeks prior to baseline endoscopy and; Are expected to remain stable for the duration of the study. and; Must be administered orally for the duration of the study. If more than one type of NSAID treatment is used, at least one type must be given orally.)
* Hp negative by UBT, serology or biopsy based test, at visit 1.

Exclusion Criteria:

* Current, or history of, gastric or duodenal ulcer
* Current, or history of, esophageal, gastric or duodenal surgery.
* History of GERD, not associated with NSAID use.
* Pain, discomfort or burning in the upper abdomen precipitated by exercise or relieved by defecation.
* Pain, discomfort or burning in the upper abdomen not associated with the use of NSAIDs, including COX-2 selective NSAIDs, as judged by the investigator.
* Endoscopic Barrett's esophagus(>3 cm) or significant dysplastic changes in the esophagus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556
Dates: Start 2000-12; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Mean change in the upper GI symptoms (pain, discomfort or
burning in the upper abdomen), rated on a 7-graded severity scale

SECONDARY OUTCOMES:
- Mean change in the upper GI symptom score
- The proportion of days with an upper GI symptom score of 'None' at 2 and 4 weeks of treatment.
- Mean upper GI symptom score by day over the duration of the study.
- Cumulative proportion of patients who achieve relief of upper GI symptoms by Week 2 and Week 4.
- Proportions of patients with upper GI symptoms during night, over the duration of the study.
- The proportion of patients with resolution or relief of investigator-recorded symptoms of heartburn, acid regurgitation, nausea & upper abdominal bloating at the 2-week, and 4-week visits.
- The mean change in the three dimensions Reflux, Abdominal pain and Indigestion of the Gastrointestinal Symptom Rating Scale (GSRS)
- Mean change in the three dimensions Emotional distress, Sleep disturbance and Food/Drink problems
- Patient's global evaluation of relief of upper GI symptom (Overall Treatment Evaluation, OTE) at the 2-week, and 4-week visits.
-Short Form-36 (SF-36) score at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (130):
- United States (32):
  - Research Site, Tallassee, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Garden Grove, California
  - Research Site, Orange, California
  - Research Site, Bradenton, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Hollywood, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tavares, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Nampa, Idaho
  - Research Site, Elkhart, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Newburgh, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Hollywood, Maryland
  - Research Site, Butte, Montana
  - Research Site, Princeton, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Endwell, New York
  - Research Site, Hewlett, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Jackson, Tennessee
  - Research Site, Pasadena, Texas
  - Research Site, Waco, Texas
  - Research Site, Edmonds, Washington
  - Research Site, Olympia, Washington
  - Research Site, Greenfield, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Australia (4):
  - Research Site, Five Dock, New South Wales
  - Research Site, Carina Heights, Queensland
  - Research Site, Kippa-Ring, Queensland
  - Research Site, Ivanhoe, Victoria
- Canada (17):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Hamilton, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sainte-Foy, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Saskatoon, Saskatchewan
  - Research Site, Quesnel
  - Research Site, St. John's
- Czechia (2):
  - Research Site, Ostrava
  - Research Site, Prague
- Italy (7):
  - Research Site, Bari, BA
  - Research Site, Genova, GE
  - Research Site, Milan, MI
  - Research Site, Perugia, PG
  - Research Site, Vicenza, VI
  - Research Site, Napoli
  - Research Site, Verona
- Norway (13):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Bærum Postterminal
  - Research Site, Gjøvik
  - Research Site, Horten
  - Research Site, Kristiansand
  - Research Site, Lillehammer
  - Research Site, Nesttun
  - Research Site, Oslo
  - Research Site, Sandvika
  - Research Site, Skien
  - Research Site, Stavanger
  - Research Site, Tromsø
- Poland (3):
  - Research Site, Bydgoszcz
  - Research Site, Sopot
  - Research Site, Warsaw
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Nové Mesto nad Váhom
- South Africa (4):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Pretoria
- Sweden (17):
  - Research Site, Bredbyn
  - Sweden, Gävle
  - Research Site, Karlskrona
  - Research Site, Kungälv
  - Research Site, Lidköping
  - Research Site, Malmo
  - Research Site, Oskarshamn
  - Research Site, Örnsköldsvik
  - Research Site, Östersund
  - Research Site, Rättvik
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Trehörningsjö
  - Research Site, Trollhättan
  - Research Site, Varberg
  - Research Site, Värnamo
  - Research Site, Västervik
- United Kingdom (29):
  - Research Site, Reading, Berks
  - Research Site, Spennymoor, Co. Durham
  - Research Site, Woking, Surrey
  - Research Site, Trowbridge, Wiltshire
  - Research Site, Ashford
  - Research Site, Audley
  - Research Site, Bath
  - Research Site, Bradford Upon Avon
  - Research Site, Chesterfield
  - Research Site, Coventry
  - Research Site, Crawley
  - Research Site, Ely
  - Research Site, Folkestone
  - Research Site, Glasgow
  - Research Site, Kilmarnock
  - Research Site, Leigh
  - Research Site, Mansfield
  - Research Site, Nottingham
  - Research Site, Pontefract
  - Research Site, Royal Tunbridge Wells
  - Research Site, Shrewsbury
  - Research Site, Stafford
  - Research Site, Swansea
  - Research Site, Trowbridge
  - Research Site, Watford
  - Research Site, Wigston
  - Research Site, Woking
  - Research Site, Worsley
  - Research Site, Yoxall